CLINICAL TRIAL: NCT00288691
Title: A Multi-center, Double-blind, Placebo-controlled, Randomized, Parallel Group Study to Evaluate the Effects of Different Doses of SH T 00127B in Women With Treatment-resistant Menorrhagia Aged 30 to 55 Years After Daily Oral Administration of Multiple Doses for 35 up to 50 Days
Brief Title: Menorrhagia Study in Women With Treatment-resistant Menorrhagia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 90955; 304667
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Menorrhagia
Keywords: Treatment-resistant menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — asoprisnil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Asoprisnil (BAY86-5294)
- Arm 2 (Experimental)
  Interventions: Drug: Asoprisnil (BAY86-5294)
- Arm 3 (Experimental)
  Interventions: Drug: Asoprisnil (BAY86-5294)
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asoprisnil (BAY86-5294) — 5mg/day
  Arms: Arm 1
Drug: Asoprisnil (BAY86-5294) — 10mg/day
  Arms: Arm 2
Drug: Asoprisnil (BAY86-5294) — 25mg/day
  Arms: Arm 3
Drug: Placebo — Placebo
  Arms: Arm 4

SUMMARY:
The aim of this study is to explore effects of the investigational product for the treatment of treatment-resistant menorrhagia without organic cause.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with treatment-resistant menorrhagia scheduled for hysterectomy.

Exclusion Criteria:

* Organic causes of menorrhagia
* Current hormone treatment

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2001-11; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Individual relative change in uterine bleeding scores by PBAC | Pretreatment cycle treatment phase

SECONDARY OUTCOMES:
Endometrial thickness | End of treatment
Adverse events collection | Whole treatment period
Bleeding pattern | Treatment period
Endometrial histology incl. immunohistochemical evaluations | End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer